CLINICAL TRIAL: NCT01245803
Title: Acute Rosuvastatin for Preventing Myocardial Damage in Patients With Acute Coronary Syndrome
Brief Title: Acute Rosuvastatin for Preventing Myocardial Damage in Patients With ACS
Acronym: AVATAR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: HYan, BeijingAnzhen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6998
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-07

CONDITIONS: Acute Coronary Syndrome; Angioplasty
Keywords: rosuvastatin; angioplasty; acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- rosuvastatin,one month,lipid lowering (Experimental): additional rosuvastatin(10mg) is given at 18hr and 4-6hr before PCI
  Interventions: Drug: additional rosuvastatin loading
- sugar pill, one month (Placebo Comparator): sugar pill is given 18-24hr and 4-6hr before PCI as control
  Interventions: Drug: placebo control

INTERVENTIONS:
Drug: additional rosuvastatin loading — additional rosuvastatin (10mg p.o.)is given at 18 hours and 4-6 hours before PCI
  Arms: rosuvastatin,one month,lipid lowering
Drug: placebo control — sugar pill is given 18-24hr and 4-6hr before PCI as control
  Arms: sugar pill, one month

SUMMARY:
Rosuvastatin reload may prevent myocardial damage in ACS patients undergoing PCI

ELIGIBILITY:
Inclusion Criteria:

* 18-75 year old
* diagnosed as acute coronary syndrome
* Plan to PCI

Exclusion Criteria:

* STEMI patient
* emergency PCI(<2h) for NSTE-ACS
* History of liver disease and myopathy (ALT/AST>3 x upper limit of normal,CK>5 x upper limit of normal)
* TG>500mg/dl,CCr<30ml/min
* inflammatory disease
* allergic to rosuvastatin
* nephrotic syndrome,hypothyroidism,systemic lupus erythematosus,myeloma,et.al.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
peri-procedural myocardial damage | 48 hours after PCI

SECONDARY OUTCOMES:
MACE | 30 days after PCI

CONTACTS AND LOCATIONS:
Locations (1):
- the 28th division, Beijing Anzhen Hospital, Beijing, Beijing Municipality, China